CLINICAL TRIAL: NCT06240390
Title: Study of the Effectiveness of Ultrasound-guided Percutaneous Neuromodulation Versus Pharmacological Treatment in Oncology Patients With Anterior Knee Pain
Brief Title: Effectiveness of Percutaneous Neuromodulation vs Pharmacological Treatment in Cancer Patients With Anterior Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Europea de Canarias (Other)
Responsible Party: Principal Investigator, Eduardo Luis Martín Javier, Master of Science Professor Eduardo Martín, Universidad Europea de Canarias
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22109-2
Record Dates: First submitted 2023-12-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Pain Cancer
Keywords: Cancer; Pain; Anterior Knee Pain; NMP
MeSH Terms: conditions — Cancer Pain; Neoplasms; Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Simple Blind, Evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epte Bipolar System 2.0 - Ultrasound-guided percutaneous neuromodulation (NMP) (Experimental): Epte Bipolar System is a medical device for health professionals that combines several techniques that extend the therapeutic variety of electrostimulation, for the treatment of different pathologies of the musculoskeletal system and peripheral and central nervous system. Ultrasound-guided percutaneous neuromodulation (NMP)
  Interventions: Device: Ultrasound-guided percutaneous neuromodulation (NMP)
- pharmacological treatment by Opioids (Experimental): Opioid analgesics are the main option for pain treatment in cancer patients, but their side effects and inadequate treatment lead to cheaper, quicker options with lower risk of addiction and/or side effects.
  Tramadol (Ultram®) Hydromorphone (Dilaudid®) Methadone (Dolophine®, Methadose®) Morphine (Apokyn®, Avinza®, Kadian®, MS-Contin®, among others) Oxycodone (OxyContin®, OxyIR®, Roxicodone®) Hydrocodone Oxymorphone (Opana®) Fentanyl (Actiq®, Duragesic®, Fentora®, Lazanda®, Subsys®, and others) Tapentadol (Nucynta®)
  Interventions: Drug: pharmacological treatment by Opioids

INTERVENTIONS:
Device: Ultrasound-guided percutaneous neuromodulation (NMP) — Epte Bipolar System is a medical device for health professionals that combines several techniques that extend the therapeutic variety of electrostimulation, for the treatment of different pathologies of the musculoskeletal system and peripheral and central nervous system. It is a nationally manufactured device that meets all quality standards, being the perfect tool for the application of techniques such as transcranial direct current stimulation. It is a versatile, compact, portable and easy to use equipment that has the ability to adapt the parameters to achieve any protocol established by scientific evidence to treat the various pathologies. The Epte® Bipolar System device has an CE Health Certificate
  Arms: Epte Bipolar System 2.0 - Ultrasound-guided percutaneous neuromodulation (NMP)
Drug: pharmacological treatment by Opioids — Opioid analgesics are the main option for pain treatment in cancer patients, but their side effects and inadequate treatment lead to cheaper, quicker options with lower risk of addiction and/or side effects.
  Other Names: pharmacological treatment - Opioids
  Arms: pharmacological treatment by Opioids

SUMMARY:
the goal of this clinical trial is to compare in cancer patients:

Is ultrasound-guided percutaneous neuromodulation useful for Anterior Knee Pain relief in cancer patients?

Participants will receive treatments of ultrasound-guided percutaneous neuromodulation and pharmacological treatment Researchers will compare ultrasound-guided percutaneous neuromodulation versus pharmacological treatment to see if Anterior Knee Pain is reduced

DETAILED DESCRIPTION:
Unhealthy lifestyles, an aging population and increased life expectancy increase the likelihood of cancer. Knee pain is one of the most common symptoms that cause functional incapacity, which requires the search and improvement of its assessment, prevention and treatment tools.

Physiotherapists are currently using ultrasound-guided Percutaneous Neuromodulation clinically. It is an easy process to perform, non-invasive, safe and economical.

Traditional therapies have been and will continue to be useful. The decrease in manufacturing costs of assessment tools such as ultrasound and neuromodulator treatment in recent years has made the acquisition of these equipment as intervention tools economical. This is because they have been shown to be useful for improving function and reducing pain.

Opioid analgesics are the main option for pain treatment in cancer patients, but their side effects and inadequate treatment lead to cheaper, quicker options with lower risk of addiction and/or side effects.

In order to improve these symptoms, it is essential to have an objective knowledge of the changes produced by neuromodulation and to be able to measure the variation of pain experienced by patients.

It has been demonstrated in recent years that assessment tools such as ultrasound and myotonometer are very useful, safe and non-invasive procedures, both have been consolidated as assessment tools that can evaluate changes and analyze the contractile properties of soft tissue quickly and safely. There are abundant literature on this subject.

Therefore, researchers suggest conducting research that improves and provides new data on the efficacy and effectiveness of treatment of ultrasound-guided percutaneous neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

The proposed inclusion criteria for the study are as follows:

* Age between 18 and 65.
* Pain in the front of the knee.
* Taking drug therapy for lower-extremity pain.
* Diagnosis of painful pathology in the anterior aspect of the knee secondary oncologic.

Exclusion Criteria:

The exclusion criteria are:

* Traumatic history
* Have had any type of analgesic treatment in the last 4 weeks (clinical, physical or orthostatic)
* No need for drug treatment within the last 30 days of study initiation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) Anterior Knee Pain changes | 12 weeks
  The Numerical Pain Rating Scale (NPRS) is a unique 11-point numeric scale that measures pain and instructs patients in clinical practice to choose a scale number from 0 to 10 with 0 for "no pain" and 10 for "worst pain possible." Its use is widely used in diseases of the knee or lower limbs, such as iliotibial girdle syndrome, sacroiliac joint dysfunction, plantar fasciitis or acute knee pain treated with microcurrents. It has also been used to treat shoulder pain in patients who have had surgery for breast cancer
Victorian Institute of Sport Assessment-Patella (VISA-P) | 12 weeks
  The VISA-P questionnaire is used for assessing the severity of symptoms in individuals with patellar tendinopathy, the term pain refers to the specific area of the patellar tendon, to mark its intensity patients should mark taking into account that 0 represents absence of pain and 10 the maximum pain imagined by the patient. In the analysis of patellar tendon pathology has already been used in repeated articles
The OKS (Oxford Knee Score) questionnaire for knee function. | 12 weeks
  The Oxford Knee Score is a well-known tool for assessing quality of life in patients with Osteo Arthritis of the knee (OA). The OKS is a self-administered questionnaire that the patient can answer in face-to-face interviews or send by mail once completed. It contains 12 questions with 5 possible answers each aimed at evaluating the perception of the quality of life of the patient in the last four weeks. Each answer receives a score of 0 to 4, where 4 is the best possible result. After the sum, you get a total score ranging from 0 to 48, where 48 is the best possible result. The Spanish adaptation of the OKS questionnaire is a reliable tool to evaluate the perception of health-related quality of life of patients with knee osteoarthritis (OA).
The Lower Limb Functional Index (LLFI). | 12 weeks
  The questionnaire contains a number of phrases (25 in total) that patients use to describe problems on their legs. Evaluating only the last few days if a phrase describes you should check that box, you can also mark it partially and if not you should leave it blank. Finally, an LLFI score is obtained where the functional index of the lower extremities is determined. The LLFI consists of 25 items with three-point response options (Yes = 1 point), ("In part" or "half" 1/2 points) and (NO Points = 0). With a gross score range of 0 to 25 points. Takes approximately 2 minutes. The score is calculated by simply adding the answers together and multiplying them by four minus 100 to convert them into a percentage scale or maximum loss of function. The LLFI questionnaire in Spanish proved to be suitable for assessing the functionality of the lower limbs and viable for the evaluation of the condition and deterioration of the lower limbs in clinical and research settings
Borg's Rating Perceived Exertion (RPE) questionnaire for perceived fatigue. | 12 weeks
  Borg created Borg's 15-point RPE scale. The modified RPE scale is 6 to 20 points. The level of physical exertion or perceived exertion is measured using the Borg 15-point RPE scale. A significant correlation was found between heart rate and Borg RPE of 15 points. In addition, this scale is believed to be a useful and cost-effective tool for monitoring exercise intensity.80 Patients in clinical practice are instructed to choose a number from the scale and assess their total effort during endurance training. A score of six indicates lack of effort, or rest, and a score of twenty indicates maximum effort, or the most exhausting exercise
Pressure pain threshold | 12 weeks
  The intensity of pain can provide relevant information, until now the measurement of pain was carried out subjectively for this reason there are efforts to develop devices to measure the intensity of painful stimuli objectively. Severity of pain also affects the patient's treatment strategy and goals because pain can cause incapacitation. Thus, several researchers have focused their efforts on creating pain-measuring devices called algometers. A pressure pain threshold (UDP) is usually used to measure this sensation. It is applied at the above point and measured in Kg/cm2.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martín, MsC, Principal Investigator — Universidad Europea de Canarias
Locations (1):
- Centro RED Tenerife, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No